CLINICAL TRIAL: NCT03301506
Title: ASSURE: An Open Label Long-Term Study to Evaluate the Safety and Tolerability of Seladelpar in Subjects With Primary Biliary Cholangitis (PBC)
Brief Title: Study of Seladelpar in Participants With Primary Biliary Cholangitis (PBC)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CB8025-31731-RE; 2020-005198-29 (EudraCT Number); 2024-511753-22-00 (EU CTIS Number)
Record Dates: First submitted 2017-09-26; First posted 2017-10-04 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Primary Biliary Cirrhosis
Keywords: PBC; Primary Biliary Cholangitis (PBC)
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — seladelpar; (2-methyl-4-(5-methyl-2-(4-trifluoromethyl-phenyl)-2H-(1,2,3)triazol-4-ylmethylsulfanyl)phenoxy)acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Seladelpar 5 mg Capsules (Experimental)
  Interventions: Drug: Seladelpar 5 mg Capsule
- Seladelpar 10 mg Capsule (Experimental)
  Interventions: Drug: Seladelpar 10 mg Capsule

INTERVENTIONS:
Drug: Seladelpar 5 mg Capsule — Participants will be assigned to a treatment group if tolerability issues noted in the previous study.
  Other Names: MBX-8025; Livdelzi®
  Arms: Seladelpar 5 mg Capsules
Drug: Seladelpar 10 mg Capsule — Participants will be assigned to a treatment group unless there are tolerability issues.
  Other Names: MBX-8025; Livdelzi®
  Arms: Seladelpar 10 mg Capsule

SUMMARY:
An Open Label Long-Term Study to Evaluate the Safety and Tolerability of Seladelpar in Subjects with Primary Biliary Cholangitis (PBC)

DETAILED DESCRIPTION:
Primary:

To evaluate the long-term safety and tolerability of seladelpar

Secondary:

* To evaluate the long-term efficacy of seladelpar
* To evaluate the effect of seladelpar on patient-reported outcomes (pruritus)

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent (signed and dated)
2. Participated in a PBC study with seladelpar
3. Females of reproductive potential must use at least one barrier contraceptive and a second effective birth control method during the study and for at least 90 days after the last dose. Male individuals who are sexually active with female partners of reproductive potential must use barrier contraception and their female partners must use a second effective birth control method during the study and for at least 90 days after the last dose

Exclusion Criteria:

Exclusion criteria are only applicable for individuals with a seladelpar interruption greater than 4 weeks prior to Day 1 of this study and for individuals who participated in CB8025-21838 irrespective of seladelpar interruption.

1. Treatment-related adverse event (AE) leading to study drug discontinuation in a previous PBC study with seladelpar
2. A medical condition, other than PBC, that in the Investigator's opinion would preclude full participation in the study or confound its results (eg, cancer, any active infection)
3. AST or ALT above 3 × the upper limit of normal (ULN)
4. Total bilirubin above 2 × ULN
5. MELD score ≥ 12. For individuals on anticoagulation medication, evaluation of the baseline INR, in concert with any current dose adjustments in anti-coagulant medications, will be taken into account when calculating this score. This will be done in consultation with the medical monitor.
6. Evidence of advanced PBC as defined by the Rotterdam criteria: albumin below 1× the lower limit of normal (LLN) AND total bilirubin above 1 × ULN)
7. eGFR ≤45 mL/min/1.73 m2 (calculated by MDRD formula)
8. Auto-immune hepatitis
9. Primary sclerosing cholangitis
10. Known history of alpha-1-antitrypsin deficiency
11. Known history of chronic viral hepatitis
12. For females, pregnancy or breast-feeding
13. Use of colchicine, methotrexate, azathioprine, or long-term use of systemic steroids (eg prednisone, prednisolone, budesonide) (>2 weeks) within 2 months prior to Screening
14. Current use of fibrates or use of fibrates within 3 months prior to Screening
15. Current use of obeticholic acid or use of obeticholic acid within 3 months prior to Screening
16. Use of an experimental or unapproved treatment for PBC within 3 months prior to Screening
17. History of malignancy diagnosed or treated, actively or within 2 years, or active evaluation for malignancy; localized treatment of squamous or non-invasive basal cell skin cancers and cervical carcinoma in-situ is allowed if appropriately treated prior to Screening
18. Treatment with any other investigational therapy or medical device within 30 days or within 5 half-lives, whatever is longer, prior to Screening
19. Any other condition(s) that would compromise the safety of the individual or compromise the quality of the clinical study, as judged by the Investigator
20. Immunosuppressant therapies (eg, cyclosporine, tacrolimus, anti-TNF or other immunosuppressive biologics)
21. Other medications that effect liver or GI functions such as absorption of medications or the roux-en-y gastric bypass procedure may be prohibited and should be discussed with the medical monitor on a case-by-case basis
22. Positive for:

    1. Hepatitis B, defined as the presence of hepatitis B surface antigen
    2. Hepatitis C, defined as the presence of hepatitis C virus ribonucleic acid (RNA)
    3. Human immunodeficiency virus (HIV) antibody
23. Active COVID-19 infection during screening

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-12-12 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent adverse events (TEAEs) (National Cancer Institute {NCI} Common Terminology Criteria for Adverse Events {CTCAE} Version 5.0), biochemistry and hematology results | Through study completion, up to 60 Months

SECONDARY OUTCOMES:
Death | 60 Months
  Occurrence of overall death
Liver transplantation | 60 Months
  Occurrence of overall liver transplantation
Change in MELD | 60 Months
  MELD score ≥ 15 for at least 2 consecutive visits
Ascites | 60 Months
  Occurrence of overall ascites requiring treatment
Hospitalization for variceal bleeding | 60 Months
  Hospitalization for new onset, or recurrence, of variceal bleeding
Hospitalization for hepatic encephalopathy | 60 Months
  Hospitalization for new onset, or recurrence, hepatic encephalopathy (as defined by a West Haven score ≥ 2)
Hospitalization for spontaneous bacterial peritonitis | 60 Months
  Hospitalization for new onset, or recurrence, spontaneous bacterial peritonitis (confirmed by culture from diagnostic paracentesis)
Response on composite endpoint | 60 Months
  Alkaline phosphate (ALP)
Response on composite endpoint | 60 Months
  Total bilirubin
Normalization of ALP | 60 Months
  Proportion of subjects with normalization of ALP
Laboratory Value: Serum Alkaline Phosphatase (ALP) | Through study completion, up to 60 Months
  Serum Alkaline Phosphatase (ALP)
Laboratory Value: Aspartate Aminotransferase (AST) | Through study completion, up to 60 Months
  Aspartate Aminotransferase (AST)
Laboratory Value: Alanine Aminotransferase (ALT) | Through study completion, up to 60 Months
  Alanine Aminotransferase (ALT)
Laboratory Value: Gamma-glutamyl Transferase (GGT) | Through study completion, up to 60 Months
  Gamma-glutamyl Transferase (GGT)
Laboratory Value: Bilirubin - Total Bilirubin | Through study completion, up to 60 Months
  Bilirubin - Total Bilirubin
Laboratory Value: Bilirubin - Conjugated Bilirubin | Through study completion, up to 60 Months
  Bilirubin - Conjugated Bilirubin
Laboratory Value: Bilirubin - Unconjugated Bilirubin | Through study completion, up to 60 Months
  Bilirubin - Unconjugated Bilirubin

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (108):
- United States (40):
  - Arkansas Diagnostic Center, Little Rock, Arkansas
  - Stanford University School of Medicine, Palo Alto, California
  - California Liver Research Institute, Pasadena, California
  - University of California Davis Medical Center, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - University of Colorado - Denver - PPDS, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Covenant Research Fort Myers, Fort Myers, Florida
  - Florida Digestive Health Specialist, Lakewood Rch, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Covenant Research, LLC, Sarasota, Florida
  - Digestive Healthcare of Georgia PC, Atlanta, Georgia
  - University of Chicago Hospitals, Chicago, Illinois
  - East Jefferson General Hospital, New Orleans, Louisiana
  - Mercy Medical Center (Baltimore), Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center - 330 Brookline Ave, Boston, Massachusetts
  - Henry Ford Health System, Novi, Michigan
  - MNGI Digestive Health PA-Plymouth, Minneapolis, Minnesota
  - Southern Therapy and Advanced Research LLC, Jackson, Mississippi
  - Saint Louis University, St Louis, Missouri
  - NYU Langone Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Rochester Medical Center - PPDS, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Northeast Clinical Research Center, LLC, Bethlehem, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Galen Medical Group, Chattanooga, Tennessee
  - Gastro One-8110 Walnut Run Rd, Cordova, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Liver Institute at Methodist Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - The Texas Liver Institute - 607 Camden St, San Antonio, Texas
  - Pinnacle Clinical Research, PLLC, San Antonio, Texas
  - Maryview Hospital Inc., d/b/a Bon Secours Liver Institute of Hampton Roads, Newport News, Virginia
  - Bon Secours Richmond Community Hospital, Inc. d/b/a Bon Secours Liver Institute of Richmond, Richmond, Virginia
  - Liver Institute Northwest, PLLC, Seattle, Washington
- Argentina (4):
  - CINME S.A. - Centro de Investigaciones Metabólicas-Viamonte 2278, Balvanera
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - DIM Clínica Privada, El Palomar
  - Hospital Italiano de La Plata, La Plata
- Australia (3):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Klinikum Wels-Grieskirchen GmbH - Standort Wels, Wels, Austria
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Canada (2):
  - University of Calgary Medicine, Calgary
  - Toronto General Hospital, Toronto
- Centro Clinico Mediterraneo, La Serena, Chile
- Fakultni nemocnice Ostrava, Ostrava, Czechia
- France (2):
  - Hospices Civils de Lyon - Hôpital de La Croix Rousse, Lyon
  - AP-HP - Hôpital Saint Antoine, Paris
- Germany (6):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitatsklinkum Erlangen-Ulmenweg 18, Erlangen
  - ifi-Institute for Interdisciplinary Medicine, Hamburg
  - Gastroenterologische Gemeinschaftspraxis Herne, Herne
  - Gastroenterologisch Hepatologisches Zentrum Kiel - Preetzer Chaussee 134, Kiel
  - Universitätsklinikum Tübingen, Tübingen
- University General Hospital of Larissa, Larissa, Greece
- Hungary (2):
  - Semmelweis Egyetem, Budapest
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz, Kaposvár
- Israel (4):
  - Carmel Medical Center, Haifa
  - Hadassah Medical Center- Ein Kerem - PPDS, Jerusalem
  - The Chaim Sheba Medical Center - PPDS, Tel Aviv
  - Tel Aviv Sourasky Medical Center Ichilov - PPDS, Tel Aviv
- Italy (3):
  - Azienda Ospedaliero-Universitaria di Modena - Ospedale Civile di Baggiovara, Modena
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone-Palermo-Piazza Delle Cliniche 2, Palermo
  - Fondazione IRCCS San Gerardo dei Tintori, Rozzano
- Mexico (2):
  - Consultorio de la Doctora Maria Sarai Gonzalez Huezo, Metepec
  - Consultorio Medico - Distrito Federal, Roma Norte
- Radboud Universitair Medisch Centrum, Nijmegen, Netherlands
- New Zealand (2):
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne Im. Prof. K. Gibinskiego Slaskiego Uniwersytetu Medycznego w Katowi, Katowice
  - ID Clinic Arkadiusz Pisula, Mysłowice
- Fundeni Clinical Institute, Bucharest, Romania
- South Korea (7):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Inje University Busan Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Songpa-Gu
- Spain (7):
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario La Paz - PPDS, Horcajo de la Sierra
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Marques de Valdecilla, Santander
- Universitätsspital Zürich, Zurich, Switzerland
- Turkey (Türkiye) (5):
  - Gazi University Faculty of Medicine, Ankara
  - Ege Universitesi Tip Fakultesi Hastanesi, Bornova
  - Ankara Bilkent City Hospital, Çankaya
  - Marmara University Pendik Training and Research Hospital, Maltepe
  - Bezmialem Vakif Universitesi Tip Fakultesi Hastanesi, Topkapı
- United Kingdom (8):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Hull Royal Infirmary, Hull
  - Barts Health NHS Trust, Royal London Hospital, Ambrose King Centre, London
  - King's College Hospital, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Queen's Medical Centre, Nottingham
  - Derriford Hospital, Plymouth
  - Queen Alexandra Hospital, Portsmouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levy C, Trivedi PJ, Kowdley KV, Gordon SC, Bowlus CL, Londono MC, Hirschfield GM, Gulamhusein A, Lawitz EJ, Vierling JM, Mayo MJ, Jacobson IM, Kremer AE, Corpechot C, Jones D, Buggisch P, Zhuo S, Proehl S, Heusner C, McWherter CA, Crittenden DB; ASSURE Investigators. Long-Term Efficacy and Safety of Selective PPARdelta Agonist Seladelpar in Primary Biliary Cholangitis: ASSURE Interim Study Results. Am J Gastroenterol. 2025 Jun 24. doi: 10.14309/ajg.0000000000003603. Online ahead of print. PMID 40553148
- [Derived] Mayo MJ, Vierling JM, Bowlus CL, Levy C, Hirschfield GM, Neff GW, Galambos MR, Gordon SC, Borg BB, Harrison SA, Thuluvath PJ, Goel A, Shiffman ML, Swain MG, Jones DEJ, Trivedi P, Kremer AE, Aspinall RJ, Sheridan DA, Dorffel Y, Yang K, Choi YJ, McWherter CA. Open-label, clinical trial extension: Two-year safety and efficacy results of seladelpar in patients with primary biliary cholangitis. Aliment Pharmacol Ther. 2024 Jan;59(2):186-200. doi: 10.1111/apt.17755. Epub 2023 Oct 30. PMID 37904314
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT03301506